CLINICAL TRIAL: NCT02716389
Title: Cervical Kinematics' Reliability: Zero Positioning Using a 3-D-bulls Eye Spirit Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SpM2016-001
Record Dates: First submitted 2016-03-04; First posted 2016-03-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Kinematics; Reliability; Cervical

ARMS (2):
- Mask on (Other)
  Interventions: Other: Zebris CMS 70; Other: 3-D Bulls Eye Spirit Meter
- Mask off (Other)
  Interventions: Other: Zebris CMS 70; Other: 3-D Bulls Eye Spirit Meter

INTERVENTIONS:
Other: Zebris CMS 70
Other: 3-D Bulls Eye Spirit Meter

SUMMARY:
The measurement of cervical spine range of motion (ROM) figures among the most common aspects of clinical diagnosis. Good reliability has been demonstrated for assessments using ultrasonic movement analysis systems, such as Zebris CMS 70 (Isny, Germany). However, in contrast to combined measurements of movement amplitudes (e.g., flexion plus extension in the sagittal plane), separating the respective components provides less reliable results. Current research suggest that this is due to the participants' determination of the zero position. This position is influenced by possible disposed treatments and, in particular, by the subject in case of subjective determination. The present study therefore aims to examine the test-retest reliability of separate ROM assessments using a bulls eye spirit meter.

Twenty healthy participants will be included in the trial that adopts a two-armed randomized, crossover design. With a washout-period of one week in between, each subject participates in two sessions in a randomised order. In both sessions, cervical ROM (flexion/extension, rotation, lateral flexion) will be measured twice (with a five-minute wait period). In all measurements, the zero position will be determined by means of a bulls eye spirit level. The difference of the two sessions consists in the design of the waiting period. In one session, the subjects will keep the mask carrying the ultrasound markers on their head. In the other session, the mask will be removed during the break.

ELIGIBILITY:
Inclusion Criteria:

* Subscribing informed consent
* Healthy

Exclusion Criteria:

* Severe orthopedic, cardiovascular, neurological, psychiatric or endocrine diseases
* Not completely healed traumata
* Drug intake in the past 48 hours
* Pregnancy
* Muscle soreness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximal cervical range of motion in flexion/extension | 2 min.

SECONDARY OUTCOMES:
Maximal cervical range of motion in lateral flexion | 2 min.
Maximal cervical range of motion in rotation | 2 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Goethe University Frankfurt/Main, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Cagnie B, Cools A, De Loose V, Cambier D, Danneels L. Reliability and normative database of the Zebris cervical range-of-motion system in healthy controls with preliminary validation in a group of patients with neck pain. J Manipulative Physiol Ther. 2007 Jul-Aug;30(6):450-5. doi: 10.1016/j.jmpt.2007.05.003. PMID 17693335